CLINICAL TRIAL: NCT00963989
Title: The START Trial: Clinical Outcome in Acute Stroke Treatment After Imaging Guided Patient Selection for Interventional Revascularization Therapy
Brief Title: Imaging Guided Patient Selection for Interventional Revascularization Therapy
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 2480.A
Record Dates: First submitted 2009-08-18; First posted 2009-08-24 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute stroke; Large cerebral vessel occlusion; Core infarct volume; Penumbra System; Revascularization; Intracerebral hemorrhage; mRS; NIHSS; Procedural serious adverse events; All cause mortality
MeSH Terms: conditions — Ischemic Stroke; Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Penumbra Device Arm (Experimental)
  Interventions: Device: Penumbra System

INTERVENTIONS:
Device: Penumbra System — The Penumbra System is used to revascularize clotted cerebral blood vessels.

SUMMARY:
The primary objective of this clinical evaluation is to determine the safety and effectiveness of the Penumbra System in a stroke cohort who presents within 8 hours from symptom and with a known core infarct volume at admission. The secondary objective is to determine if there is a correlation between infarct volume and functional outcome in treated patients at 90 days post-procedure.

DETAILED DESCRIPTION:
Study Title: The START Trial: Clinical Outcome in Acute Stroke Treatment after Imaging Guided Patient Selection for Interventional Revascularization Therapy

Study Objective: The objective of this clinical evaluation is to determine the safety and effectiveness of the Penumbra System in a stroke cohort who presents within 8 hours from symptom onset and with a known core infarct volume at admission. The data will also be used to determine if there is a correlation between infarct volume and functional outcome at 90 days post-procedure. Safety is defined by the procedural serious adverse events, and effectiveness is defined by the rate of revascularization (TIMI 2-3/TICI 2a-3) and good functional outcome. Good functional outcome is defined by a modified Rankin scale (mRS) score of 2 or less at 90 days post-procedure. Core infarct volume at admission will be assessed by computed tomography perfusion (CTP), computed tomography angiography (CTA) or magnetic resonance DWI scans. The core infarct volumes will be sub-grouped by <50cc, 50-100cc and >100cc to determine the correlation with patient functional outcome.

Study Design: A prospective, single arm, multi-center trial. Up to 200 patients at up to 45 centers will be enrolled in the study. It is anticipated that up to 150 evaluable patients will be needed for analysis.

Patient Population: Patients presenting with symptoms of acute ischemic stroke within 8 hours from symptom onset and with a known imaging-defined infarct volume will be enrolled for interventional treatment by the Penumbra System to achieve revascularization of the target vessel territory.

Indication: The Penumbra System is intended for use in the revascularization of patients with acute ischemic stroke secondary to intracranial large vessel occlusive disease (within the internal carotid, middle cerebral - M1 and M2 segments, basilar, and vertebral arteries) within 8 hours of symptom onset.

Sample Size Justification: Up to 200 subjects will be enrolled in order to obtain up to 150 evaluable patients. Assuming a post-procedure angiographic success (TIMI 2-3/TICI 2a-3) rate of 80% (120/150), the expected two-sided exact binomial 95% confidence interval is (72.7%, 86.1%). Assuming a 90-day mRS success (mRS 0-2) rate of 30%, the expected two-sided exact binomial 95% confidence interval is (22.8%, 38.0%). Additionally, the study results will be used for sample size estimates for a potential future randomized, concurrent controlled trial.

Core Laboratory and Clinical Event Committee An independent Core Lab will review and score all imaging scans for infarct volume, TIMI, TICI and ICH. A Clinical Event Committee will adjudicate all Serious Adverse Events for severity and causality (disease-, procedure-, drug-, or device-relatedness.

Study Rationale: Use of interventional revascularization techniques offer several potential clinical benefits by improving cerebral perfusion to the target vascular territory in certain patients. The validation of a simple, pragmatic, and executable image guided patient selection paradigm may identify a cohort of acute stroke patients who will benefit from interventional treatment by the Penumbra System and in whom revascularization as a treatment for acute stroke will be indicated.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 85 years of age.
* Evidence of proximal anterior circulation large vessel occlusion (TIMI /TICI 0-1) (Tables 2A & B). Target vessel occlusion may include the supra-clinoid segment of the ICA through the M1 segment of the MCA.
* Presented with symptoms consistent with acute ischemic stroke within 8 hours of symptom onset. Patients who presented within 3 hours must be ineligible or refractory to IV rtPA therapy.
* At time of enrollment, neurological deficit resulting in an NIH Stroke Scale (NIHSS) score of 10 or greater.
* Core infarct volume assessed by CTP, CTA or DWI scans within 60 minutes to arterial puncture.
* Signed informed consent.

Exclusion Criteria:

* History of stroke in the past 3 months.
* Vessel tortuosity too difficult to allow endovascular access.
* Pre-existing neurological or psychiatric disease that could confound the study results such as a pre-stroke mRS score of 1 or greater.
* Known severe allergy to contrast media.
* Uncontrolled hypertension (defined as systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg).
* Noncontrast CT evidence of the following conditions before enrollment:

  * Significant mass effect with midline shift;
  * Evidence of intracranial hemorrhage.
* Angiographic evidence of an arterial stenosis proximal to the occlusion that could prevent thrombus removal.
* Angiographic evidence of preexisting arterial injury.
* Life expectancy less than 90 days.
* Participation in another clinical investigation that could confound the evaluation of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siu P Sit, PhD, Study Director — Penumbra Inc.
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Penumbra Device Arm
Started | 146
Completed | 127
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Penumbra Device Arm
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 64
Baseline NIHSS [Mean (Inter-Quartile Range); unit: units on a scale] — National Institutes of Health Stroke Scale ranges from 0-42, with higher scores being worse.
  units on a scale | 19 [14 to 23]

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcome as Defined by a mRS of 0-2 at 90 Days Post-procedure
Description: Modified Rankin Scale (mRS) ranges from 0 to 5, with higher scores being worse.
Time Frame: At 90 days post-procedure
Population: 16 subjects with missing 90-day mRS assessment and 3 withdrew consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Device Arm
Number analyzed (Participants) | 127
Participants | 57

2. Primary Outcome: Angiographic Assessment of Vessel Patency as Measured by TIMI Score
Description: Defined by Number of participants with Thrombolysis in Myocardial Infarction (TIMI) 2-3.
  A lower score means a worse outcome and higher scores means better outcome on a scale of 0-3.
Time Frame: At immediate post-procedure
Population: One subject had two sites of occlusion
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Device Arm
Number analyzed (Participants) | 147
Participants | 122

3. Primary Outcome: Angiographic Assessment of Vessel Patency as Measured by Modified TICI Score
Description: Defined by number of participants with modified thrombolysis in cerebral infarction (TICI) 2-3.
  A lower score means a worse outcome and higher scores means better outcome on a scale of 0-3.
Time Frame: At immediate post-procedure
Population: One subject had two sites of occlusion
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Device Arm
Number analyzed (Participants) | 147
Participants | 122

4. Primary Outcome: Procedural Serious Adverse Events During the Procedure
Description: Defined by serious adverse events (SAEs) within 24 hours of the procedure
Time Frame: During the procedure, approximately 24 hours
Measure: Number; unit: events
Arm/Group | Penumbra Device Arm
Number analyzed (Participants) | 146
events | 40

5. Secondary Outcome: Good Neurological Recovery Post-procedure as Defined by a 10 Points or More Improvement on the NIHSS at Discharge
Time Frame: At Discharge, an average of 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Device Arm
Number analyzed (Participants) | 112
Participants | 47

6. Secondary Outcome: Incidence of Symptomatic and Asymptomatic Hemorrhage Based on the ECASS Criteria and Patient Neurological Status Within 24 Hours of the Procedure
Time Frame: Within 24 hours of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Device Arm
Number analyzed (Participants) | 146
Participants | 18

7. Secondary Outcome: All Cause Mortality at 90 Days Post-procedure
Time Frame: At 90 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra Device Arm
Number analyzed (Participants) | 146
Participants | 37

ADVERSE EVENTS:
Arm/Group | Penumbra Device Arm
All-Cause Mortality (participants affected / at risk) | 37/146
Serious Adverse Events (participants affected / at risk) | 8/146
Other Adverse Events (participants affected / at risk) | 14/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Penumbra Device Arm (N=146)
Carotid artery dissection (Nervous system disorders) | 1
Cerebral artery occlusion (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral vasoconstriction (Nervous system disorders) | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1
Vessel perforation (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Penumbra Device Arm (N=146)
Infusion site extravasation (General disorders) | 1
Cerebral artery embolism (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral vasoconstriction (Nervous system disorders) | 7
Haemorrhagic transformation stroke (Nervous system disorders) | 1
Vascular dissection (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No